CLINICAL TRIAL: NCT04250025
Title: A Prospective Randomized, Open-label, Blind Evaluator, Evaluating the Efficacy of Proximal Venous Angioplasty-stenting vs Optimal Medical Treatment on Post-thrombotic Syndrome Reduction
Brief Title: Angioplasty-stenting vs Optimal Medical Treatment on Post-thrombotic Syndrome Reduction
Acronym: EndoPTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A01311-56
Record Dates: First submitted 2020-01-27; First posted 2020-01-31 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-02

CONDITIONS: Post Thrombotic Syndrome
MeSH Terms: conditions — Postthrombotic Syndrome

STUDY DESIGN:
Intervention Model Description: Patients are randomised into two groups:Experimental Group: 60 patients benefit from immediate venous angioplasty stenting plus medical treatment, i.e. elastic compression and anticoagulation Control Group: 60 patients benefit from standard treatment for 6 months i.e elastic compression and anticoagulation if needed. Notably, if patients were no longer on anticoagulant treatment at the time of screening and inclusion, this treatment will not be reintroduced.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUPE (Experimental): 60 patients benefit from immediate venous angioplasty stenting plus medical treatment, i.e. elastic compression and anticoagulation
  Interventions: Procedure: 60 patients benefit from immediate venous angioplasty stenting plus medical treatment, i.e. elastic compression and anticoagulation
- CONTRO GROUPE (No Intervention): 60 patients benefit from standard treatment for 6 months i.e elastic compression and anticoagulation if needed. Notably, if patients were no longer on anticoagulant treatment at the time of screening and inclusion, this treatment will not be reintroduced.

INTERVENTIONS:
Procedure: 60 patients benefit from immediate venous angioplasty stenting plus medical treatment, i.e. elastic compression and anticoagulation — 60 patients benefit from immediate venous angioplasty stenting plus medical treatment, i.e. elastic compression and anticoagulation
  Arms: EXPERIMENTAL GROUPE

SUMMARY:
The project will highlight the potential benefit of endovascular therapy on post thrombotic syndrome reduction after proximal iliac DVT. There is actually not real standard of care for the treatment of this pathology. A clear evidence of efficacy of endovascular therapy will be of great benefit for both the patients and the healthcare system, and will provide new data for further international guidelines

DETAILED DESCRIPTION:
Benefit(s) for the individual:

Patients included in the experimental arm of the study will attempt to a strong reduction of PTS. In addition, all patients of the study will benefit from a careful follow-up thanks to the availability of physicians involved in the study, optimization of quality of compression therapy and anticoagulant treatment, and will be strongly encouraged to regular physical activity.

Group(s) Benefits:

About 100 000 to 150 000 persons develop VTE each year in France, among which about 5% will develop severe and disabling PTS. Validation of interventional therapy may provide a major clinical improvement for these patients in terms of morbidity and quality of life. The economic impact is likely to be improved.

Risk(s) to the individual(s)

The first risk is related to interventional treatment, i.e. haemorrhages or early DVT recurrence. The use of endovascular approach will reduce the haemorrhagic risk compared to open surgery, and the risk of recurrence will be controlled by anticoagulant.

The second risk is related to antithrombotic treatment, i.e. combination of aspirin plus anticoagulant, then anticoagulant alone. The combined therapy will be used during a short one-month treatment reducing the risk, and the patients are already trained to anticoagulant treatment. Moreover, it is attempted, regarding the characteristics of patients eligible to interventional procedure that these patients are at low risk of bleeding.

2.3.2 Benefit/risk balance

The benefit/risk balance will be positive.

Patients included in the experimental arm of the study will attempt to a strong reduction of PTS, although the procedure is mastered with limited risk. The fact that investigators already practice this procedure in everyday practice contributes to reducing this risk.

Patients included in the control group will be treated according to the current clinical practice and national and international recommendations. In case of non-resolution of symptoms, they will be invited to interventional procedure 6 months later.

In addition, all patients of the study will benefit from a careful follow-up.

Adverse events will be supervised to control the benefit/risk balance between the two arms. Moreover, the choice to propose a delayed endovascular procedure for control group's patients is primordial because even if the medical treatment is the current clinical practice and national and international recommendations, endovascular procedure has emerged like key treatment. So, to avoid the risk that patients refuse study or leave the study if they are randomized in medical treatment, we propose a 6 months delayed intervention for these patients. This delay of 6 months is reasonable for the adherence of patients to the study.

With these patients, we will have access to results of endovascular procedure at 6 months after delayed intervention, increasing the pool of data on the effect of endovascular procedure.

2.4 Expected Impact

The project will highlight the potential benefit of endovascular therapy on post thrombotic syndrome reduction after proximal iliac DVT. There is actually not real standard of care for the treatment of this pathology. A clear evidence of efficacy of endovascular therapy will be of great benefit for both the patients and the healthcare system, and will provide new data for further international guidelines

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years' old
* Patient with disabling PTS defined as a Villalta score ≥ 10, more than 6 months after unilateral proximal deep vein thrombosis (first or recurrent episode) involving at least iliac vein. A contralateral distal or superficial vein thrombosis was not considered as bilateral thrombosis.

Rational for main inclusion criteria:

Patients would be screened more than 6 months after the index DVT event to be sure that symptoms were related to chronic phase of PTS and not to the acute DVT event.

Although endovascular therapy has actually matured to propose a systematic evaluation, the procedure remains experimental with potential risks. Therefore, the study must focus on patients with advanced PTS and iliofemoral obstruction, since this population appears to have the greatest attempted benefit.

Exclusion Criteria:

* Index DVT without iliac thrombosis
* Bilateral proximal deep vein thrombosis or Inferior vena cava thrombosis
* Lower limb arteriopathy defined as ante-brachial index < 0.5
* Vena cava filter
* Venous ulcers ≥ 50 cm²
* Life expectancy < 6 months
* Contraindication to anticoagulant treatment by direct oral anticoagulant
* Contraindication to the use of low-dose aspirin (100 mg)
* Use of dual antiplatelet agents aspirin/clopidogrel
* Use of Prasugrel or Ticagrelor
* Previous venous recanalization of the same leg
* Impossible to follow-up
* Contraindication to contrast iodine
* Renal insufficiency (Cockroft <30 ml/min, (less than 3 months old))
* Subject in exclusion period from another study,
* Pregnant or breastfeeding women
* Subject under administrative or judicial control
* Subject under legal protection
* Subject hospitalized for psychiatric care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of percentage of patients with corrected PTS (Villalta< 5 i.e. absence of PTS) at 6 months after randomization in control group and 6 months after intervention in experimental group. | 6 months
  Comparison of percentage of patients with corrected PTS (Villalta< 5 i.e. absence of PTS) at 6 months after randomization in control group and 6 months after intervention in experimental group.

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble-Alps University Hospital (CHUGA), Grenoble, CS 10217, France

REFERENCES:
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829